CLINICAL TRIAL: NCT00403065
Title: Quality of Life After Radiotherapy & Steroids. A Phase III Multi-Centre Randomised Controlled Trial to Assess Whether Optimal Supportive Care Alone (Including Dexamathasone) is As Effective as Optimal Supportive Care (Including Dexamethasone ) Plus Whole Brain Radiotherapy in the Treatment of Patients With Inoperable Brain Metastases From Non-Small Cell Lung Cancer
Brief Title: Dexamethasone and Supportive Care With or Without Whole-Brain Radiation Therapy in Treating Patients With Non-Small Cell Lung Cancer That Has Spread to the Brain and Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical Research Council (Other Government)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000517194; MRC-LU24-QUARTZ; EU-20653; ISRCTN3826061; TROG 07.02
Record Dates: First submitted 2006-11-21; First posted 2006-11-23 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2007-01

CONDITIONS: Lung Cancer; Metastatic Cancer
Keywords: recurrent non-small cell lung cancer; stage IV non-small cell lung cancer; tumors metastatic to brain
MeSH Terms: conditions — Lung Neoplasms; Neoplasm Metastasis; Carcinoma, Non-Small-Cell Lung; Brain Neoplasms | interventions — Dexamethasone; Radiotherapy

INTERVENTIONS:
Drug: dexamethasone
Procedure: quality-of-life assessment
Radiation: radiation therapy

SUMMARY:
RATIONALE: Steroid therapy, such as dexamethasone, may reduce swelling, pain, and other symptoms of inflammation and may be effective in treating some of the problems caused by cancer and cancer treatment. Supportive care improves the quality of life of patients with a serious or life-threatening disease, and prevents or treats symptoms of cancer, side effects of treatment, and other problems related to cancer or its treatment. Radiation therapy uses high-energy x-rays to kill tumor cells. It is not yet known whether dexamethasone given together with supportive care is more effective with or without whole-brain radiation therapy in treating patients with brain metastases.

PURPOSE: This randomized phase III trial is studying dexamethasone and supportive care to see how well it works with or without whole-brain radiation therapy in improving the quality of life of patients with non-small cell lung cancer that has spread to the brain and cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the efficacy of dexamethasone with vs without whole-brain radiotherapy in combination with optimal supportive care, in terms of patient assessed quality adjusted life years, in patients with inoperable brain metastases secondary to non-small cell lung cancer.

Secondary

* Compare the overall survival of patients treated with these regimens.
* Assess the Karnofsky performance status of patients treated with these regimens.
* Assess the symptoms of patients treated with these regimens.
* Determine the feasibility of assessing and measuring caregiver concerns.

OUTLINE: This is a randomized, controlled, multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I (experimental): Patients receive dexamethasone*. Patients receive optimal supportive care (OSC) including a prescription of a proton pump inhibitor while on dexamethasone, parallel nursing support, access to additional specialists (e.g., pain-relief service, palliative care team, medical social worker, or physiotherapist), and open access to follow-up in a specialist clinic. OSC may also include analgesics, bronchodilators, and other supportive treatment as needed.
* Arm II (control): Patients receive dexamethasone* and OSC as in arm I. Patients also undergo whole-brain radiotherapy once daily for 5 days in the absence of disease progression or unacceptable toxicity.

NOTE: *Patients who are receiving prednisolone at randomization need to convert to dexamethasone immediately.

All patients undergo telephone assessment, including quality of life assessment, once a week for 12 weeks and then once every 4 weeks thereafter. Consenting caregivers complete questionnaire over the telephone once a week to assess the impact of the patient's disease and treatment on the caregiver's quality of life.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: At least 1,000 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed primary non-small cell lung cancer
* Must have brain metastases confirmed by CT scan or MRI

  * Unresectable disease OR surgery is deemed inappropriate
* The benefit or lack of benefit of whole-brain radiotherapy (WBRT) cannot be clearly defined

  * Any known certainty of the benefit or lack of benefit of WBRT is not allowed

PATIENT CHARACTERISTICS:

* No prior or concurrent uncontrolled illness that could preclude study treatment or comparisons
* Must be able to respond to weekly telephone assessment questions

PRIOR CONCURRENT THERAPY:

* More than 1 week since prior epidermal growth factor receptor inhibitors
* More than 1 month since prior chemotherapy
* More than 1 month since prior surgery for brain metastases
* No prior radiotherapy to the brain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2006-10; Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Patient-assessed quality adjusted life years

SECONDARY OUTCOMES:
Overall survival
Karnofsky performance status
Patient symptoms
Assessment and measurement of caregiver concerns

CONTACTS AND LOCATIONS:
Overall Officials: Paula Mulvenna, Study Chair — Northern Centre for Cancer Treatment at Newcastle General Hospital
Locations (70):
- United Kingdom (70):
  - Wansbeck General Hospital, Ashington, England
  - Sussex Cancer Centre at Royal Sussex County Hospital, Brighton, England
  - Bristol Haematology and Oncology Centre, Bristol, England
  - Addenbrooke's Hospital, Cambridge, England
  - Papworth Hospital, Cambridge, England
  - Cumberland Infirmary, Carlisle, England
  - Gloucestershire Oncology Centre at Cheltenham General Hospital, Cheltenham, England
  - Saint Richards Hospital, Chichester, England
  - Castle Hill Hospital, Cottingham, England
  - Walsgrave Hospital, Coventry, England
  - Darlington Memorial, Darlington, England
  - Derbyshire Royal Infirmary, Derby, England
  - Dorset County Hospital, Dorchester, England
  - University Hospital of North Durham, Durham, England
  - Bishop Auckland Hospital, Durham, England
  - Royal Devon and Exeter Hospital, Exeter, England
  - Queen Elizabeth Hospital, Gateshead, England
  - Diana Princess of Wales Hospital, Grimsby, England
  - Hereford Hospitals, Hereford, England
  - Huddersfield Royal Infirmary, Huddersfield, West Yorks, England
  - Princess Royal Hospital at Hull and East Yorkshire NHS Trust, Hull, England
  - Ipswich Hospital, Ipswich, England
  - Queen Elizabeth Hospital, Kings Lynn, England
  - Cookridge Hospital, Leeds, England
  - Aintree University Hospital, Liverpool, England
  - Whipps Cross Hospital, London, England
  - Newham University Hospital, London, England
  - Homerton University Hospital, London, England
  - Saint Bartholomew's Hospital, London, England
  - Guy's Hospital, London, England
  - St. Mary's Hospital, London, England
  - UCL Cancer Institute, London, England
  - Christie Hospital, Manchester, England
  - Clatterbridge Centre for Oncology, Merseyside, England
  - James Cook University Hospital, Middlesbrough, England
  - Northern Centre for Cancer Treatment at Newcastle General Hospital, Newcastle upon Tyne, England
  - North Tyneside Hospital, North Shields, England
  - Friarage Hospital, North Yorks, England
  - Northampton General Hospital, Northampton, England
  - Mount Vernon Cancer Centre at Mount Vernon Hospital, Northwood, England
  - Nottingham City Hospital, Nottingham, England
  - George Eliot Hospital, Nuneaton, England
  - Dorset Cancer Centre, Poole Dorset, England
  - Portsmouth Oncology Centre at Saint Mary's Hospital, Portsmouth Hants, England
  - Whiston Hospital, Prescot Merseyside, England
  - Berkshire Cancer Centre at Royal Berkshire Hospital, Reading, England
  - Alexandra Healthcare NHS, Redditch, Worcestershire, England
  - South Tyneside District Hospital, South Shields, England
  - Southampton General Hospital, Southampton, England
  - Southport and Formby District General Hospital, Southport, England
  - University Hospital of North Tees, Stockton-on-Tees, England
  - Taunton and Somerset Hospital, Taunton, England
  - Torbay Hospital, Torquay, England
  - Royal Cornwall Hospital, Truro, England
  - Walsall Manor Hospital, Walsall, England
  - South Warwickshire Hospital, Warwick, Warwickshire, England
  - New Cross Hospital, Wolverhampton, England
  - Worcester Royal Hospital, Worcester, England
  - Cancer Care Centre at York Hospital, York, England
  - Centre for Cancer Research and Cell Biology at Queen's University Belfast, Belfast, Northern Ireland
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Ninewells Hospital, Dundee, Scotland
  - Hairmyres Hospital, East Kilbride, Scotland
  - Edinburgh Cancer Centre at Western General Hospital, Edinburgh, Scotland
  - Beatson West of Scotland Cancer Centre, Glasgow, Scotland
  - Raigmore Hospital, Inverness, Scotland
  - Crosshouse Hospital, Kilmarnock, Scotland
  - Velindre Cancer Center at Velindre Hospital, Cardiff, Wales
  - Llandough Hospital, Llandough, Wales
  - Glan Clwyd Hospital, Rhyl, Denbighshire, Wales